CLINICAL TRIAL: NCT00055913
Title: A Phase I/II Study Of Bevacizumab (rhuMAb VEGF) In Combination With OSI-774 For Patients With Recurrent Or Metastatic Cancer Of The Head And Neck
Brief Title: Bevacizumab and Erlotinib in Treating Patients With Recurrent or Metastatic Head and Neck Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02520; NCI-2012-02520 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000271444; UCCRC-NCI-5701; UCCRC-11956A; NCI-5701; 11956A (Other: University of Chicago); 5701 (Other: CTEP); P30CA014599 (NIH); N01CM62201 (NIH)
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Salivary Gland Squamous Cell Carcinoma; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Larynx; Stage IV Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IV Squamous Cell Carcinoma of the Oropharynx; Stage IV Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Bevacizumab; Erlotinib Hydrochloride

ARMS (2):
- Arm I (Experimental): Patients receive bevacizumab IV over 30-90 minutes on day 15 and oral erlotinib on days 1-28. All subsequent courses patients receive oral erlotinib on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Drug: erlotinib hydrochloride; Other: laboratory biomarker analysis
- Arm II (Experimental): Patients receive bevacizumab IV over 30-90 minutes on day 1 and oral erlotinib on days 1-28. All subsequent courses patients receive oral erlotinib on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Drug: erlotinib hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Drug: erlotinib hydrochloride — Given orally
  Other Names: CP-358,774; erlotinib; OSI-774
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase I/II trial is to see if combining erlotinib with bevacizumab works better in treating patients who have recurrent or metastatic head and neck cancer. Erlotinib may stop the growth of tumor cells by blocking the enzymes needed for tumor cell growth. Monoclonal antibodies, such as bevacizumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or deliver cancer-killing substances to them. Combining erlotinib with bevacizumab may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose and dose-limiting toxicity of bevacizumab when administered with erlotinib in patients with recurrent or metastatic head and neck cancer.

II. Determine the objective response rate and stable disease/absence of early progression in patients treated with this regimen.

OUTLINE: This is a dose-escalation study of bevacizumab followed by a randomized, multicenter study.

Phase I: Patients receive bevacizumab IV over 30-90 minutes on day 1 and oral erlotinib on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of bevacizumab until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Phase II: Course 1 is 28 days in length. All subsequent courses are 21 days.

Course 1: Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive bevacizumab IV over 30-90 minutes on day 15 and oral erlotinib on days 1-28.

Arm II: Patients receive bevacizumab IV over 30-90 minutes on day 1 and oral erlotinib on days 1-28.

All subsequent courses: All patients receive bevacizumab as in arm II and oral erlotinib on days 1-21.

Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed squamous cell cancer of the head and neck

  * Recurrent or metastatic disease
  * Determined to be incurable by surgery or radiotherapy
* Measurable disease
* No tumor involvement encasing or too close in proximity to a major artery or vein
* No known brain metastases
* No prior or concurrent CNS disease
* No primary brain tumor
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* More than 12 weeks
* No history of bleeding diathesis
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* INR less than 1.5
* Bilirubin normal
* AST and ALT no greater than 2.5 times upper limit of normal
* Creatinine normal
* Creatinine clearance at least 60 mL/min
* No significant renal impairment
* 24-hour urinary protein less than 0.5 g required if more than trace proteinuria at baseline
* No uncontrolled hypertension
* No symptomatic congestive heart failure
* No serious cardiac arrhythmia requiring medication
* No deep venous thrombosis
* No prior stroke
* No New York Heart Association class II-IV heart disease
* No grade II-IV peripheral vascular disease within the past year
* No arterial thromboembolic event within the past 6 months, including any of the following:

  * Unstable angina pectoris
  * Myocardial infarction
  * Transient ischemic attack
  * Cerebrovascular accident
* No clinically significant peripheral artery disease
* No significant ophthalmologic abnormalities* including any of the following:

  * Severe dry eye syndrome
  * Keratoconjunctivitis sicca
  * Sjögren's syndrome
  * Severe exposure keratopathy
  * Disorders that might increase the risk for epithelium-related complications (e.g., bullous keratopathy, aniridia, severe chemical burns, neutrophilic keratitis)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior allergic reactions to compounds of similar chemical or biologic composition to bevacizumab or other study agents
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* No significant traumatic injury within the past 28 days
* No other concurrent uncontrolled illness
* No psychiatric illness or social situation that would preclude study compliance
* No ongoing or active infection requiring parenteral antibiotics
* No serious non-healing wound ulcer or bone fracture
* No seizures not controlled by standard medical therapy
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* More than 4 weeks since prior radiotherapy
* More than 4 weeks since prior major surgery
* More than 4 weeks since prior open biopsy
* Recovered from prior therapy
* No more than 1 prior regimen for recurrent disease
* No prior epidermal growth factor receptor (EGFR)-based therapy for recurrent disease
* No prior vascular EGFR-based therapy for recurrent disease
* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent chronic use of aspirin (325 mg/day or more) or other nonsteroidal anti-inflammatory drugs
* No concurrent warfarin or heparin, including low-molecular weight heparin
* No other concurrent or recent (within 1 month) thrombolytic agents or full-dose anticoagulants (except to maintain patency of preexisting, permanent indwelling IV catheters)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2003-03; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of bevacizumab when used in combination with erlotinib hydrochloride determined by dose-limiting toxicities (Phase I) | 28 days
Objective response rate (CR + PR) evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) (Phase II) | Up to 6 months
Progression-free survival rate (Phase II) | Time from the start of treatment until disease progression or death, assessed up to 7 years
Overall survival rate (Phase II) | Up to 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Tanguy Seiwert, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Cohen EE, Davis DW, Karrison TG, Seiwert TY, Wong SJ, Nattam S, Kozloff MF, Clark JI, Yan DH, Liu W, Pierce C, Dancey JE, Stenson K, Blair E, Dekker A, Vokes EE. Erlotinib and bevacizumab in patients with recurrent or metastatic squamous-cell carcinoma of the head and neck: a phase I/II study. Lancet Oncol. 2009 Mar;10(3):247-57. doi: 10.1016/S1470-2045(09)70002-6. Epub 2009 Feb 7. PMID 19201650